CLINICAL TRIAL: NCT00199732
Title: Evaluation of cccDNA and Total HBV DNA Kinetics in Lymphocytes, Total Blood and Serum in Chronic Hepatitis B Patients Treated With Adefovir Dipivoxil and Peg Interferon Alpha 2a
Acronym: DNA-EVAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: I04002
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; CCC DNA kinetics; Total HBV DNA kinetics; Adefovir-Dipovixil; Peg interferon alpha 2a
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Serum HBV DNA is a referent but insufficient marker of therapeutic follow-up in chronic hepatitis B treatment. Intra hepatic cccDNA disappearance reflects HBV eradication in the liver.

Intra lymphocyte cccDNA could be a new marker of HBV eradication after treatment.

The major interest of this marker is that it can be measured by a simple blood test instead of a liver biopsy.

DETAILED DESCRIPTION:
- Studying intra lymphocyte and blood cccDNA: before inclusions, D0 then each month during the first three months each three months during treatment and follow-up.

- Viral kinetics:Before inclusions, at D0, then monthly till the end of treatment and follow-up: Evolution of quantitative viraemia in serum Evolution of quantitative viraemia in circulating lymphocytes Evolution of quantitative viraemia in total blood

- Studying viral genotypes

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >18 years of age and <70 years of age
* Patients AgHbs+ and AgHbe+ or AgHbe-, and B viral DNA >104 copies/ml PCR COBAS MONITOR
* Patients treated with adefovir dipivoxil and peg interferon alpha 2a
* Chronic liver disease consistent with chronic hepatitis B infection on a biopsy obtained within the past 24 months
* Naïve patients or patients having a relapse or a therapeutic failure after monotherapy lamivudine or interferon, or bitherapy interferon alpha-lamivudine

Exclusion Criteria:

* Co-infection HIV, HCV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B infection and treated with adefovir dipivoxil and peg interferon alpha 2a.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Kinetic cccDNA | 6 months
  Studying the kinetics of cccDNA in cells and whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Loustaud-Ratti, MD, Principal Investigator — University Hospital, Limoges
Locations (4):
- France (4):
  - Service d'Hépato-gastroentérologie, Limoges
  - Service de Médecine Interne, Limoges
  - Service de Virologie, Limoges
  - Service des Maladies Infectieuses et Tropicales, Limoges